CLINICAL TRIAL: NCT06812611
Title: Effects of High Intensity Laser Therapy In Lower Limb Muscle Injuries: a Randomized Controlled Study
Brief Title: Effects of High Intensity Laser Therapy in Muscle Injuries
Acronym: THEALinMJ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THEALinMJ
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-01

CONDITIONS: Muscle Tear
Keywords: laser; high energy; limb; muscle tear
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Energy Laser Group (Experimental): The multimodal high energy laser therapy treatment with thermal control (THEAL) will be delivered with an Ixyon XP device (Mectronic, Bergamo, Italy) which allows the delivery of 4 wavelengths (650 nm, 810 nm, 980 nm and 1064 nm), with continuous and pulsed mode, average power up to 30 W, administering 10 sessions every other day. The patients will simultaneously carry out the rehabilitation treatment exercises, as was expected in the control group.
  Interventions: Device: High Energy Laser Group; Other: Exercise
- Exercise Group (Active Comparator): All patients will receive a rehabilitation protocol of 5 weekly sessions lasting approximately 60 minutes, for approximately 3 weeks. During the early post-injury phases, the protocol will include isometric exercises to strengthen core stability. These exercises will each be performed for 3 sets of 30 seconds, although the number of sets and repetitions may vary depending on the athlete's response.
  Interventions: Other: Exercise

INTERVENTIONS:
Device: High Energy Laser Group — The multimodal high energy laser therapy treatment with thermal control (THEAL) will be delivered with an Ixyon XP device (Mectronic, Bergamo, Italy) which allows the delivery of 4 wavelengths (650 nm, 810 nm, 980 nm and 1064 nm), with continuous and pulsed mode, average power up to 30 W, administering 10 sessions every other day.
  The patients will simultaneously carry out the rehabilitation treatment exercises, as was expected in the control group.
  Arms: High Energy Laser Group
Other: Exercise — Daily exercise

SUMMARY:
Muscle injuries are frequent traumatic events in daily life, particularly during sports. In sports, their incidence varies from 10% to 55% of total injuries. According to the Mueller Wohlfart classification, muscle injuries are classified into direct traumatic injuries (contusion-laceration) and indirect traumatic injuries, which are further divided into non-structural injuries (grade I and II) and structural injuries. Structural lesions are further divided into partial muscle lesions (grade III): 3 A, minor partial lesion, i.e. lesion of one or more primary bundles with a secondary bundle; 3 B, moderate partial lesion, i.e. lesion of at least one secondary bundle and with a rupture area < 50% of the muscle surface; and (sub)total muscle injury (grade IV).

DETAILED DESCRIPTION:
In the acute phase, the current management of muscle injuries is essentially based on the PRICE protocol (protection, rest, ice, compression, elevation), although there are still no randomized clinical trials in the literature demonstrating its real effectiveness. Subsequently, the player undertakes rehabilitation with exercises and therapies aimed at resolving the edema, repairing the injury, strengthening the muscles and restoring athletic movements.

Biostimulations (laser therapy, diathermy, US, etc) are applied in muscle lesions for their analgesic and anti-inflammatory action, but to date there is a lack of adequate clinical evidence. The high energy laser has a great penetration force deep into the tissues and through its photochemical effects, increases mitochondrial oxidation and facilitates the formation of adenosine triphosphate (ATP), as well as inducing an increase in metabolism and blood circulation, with rapid absorption of edema and elimination of exudates. This induces an important biological action, causing muscle relaxation and inhibition of free nerve endings resulting in an immediate reduction in pain.

Preclinical studies have shown that physical therapies, such as high-energy laser therapy, improve muscle regeneration. On the other hand, to date few clinical studies have investigated the effects of biostimulations on muscle injuries. Medeiros et al. did not find benefits in the application of low energy laser in the treatment of muscle injuries, hypothesizing that a late application may have undermined the effects of biostimulation, which is fundamental in the first days of a late injury. Scaturro et al. , applying a combination of high energy laser and diathermy in association with rehabilitation treatment within 5 days of muscle injury, found positive effects on pain remission, return to sporting activity and the number of relapses. On the other hand, in this study, the contextual administration of two biostimulations (high energy laser and tecar therapy) does not allow us to discriminate the biological and clinical effects attributable to each of the two therapeutic methods.

Therefore, the aim of the present study is to investigate the effects of high intensity laser therapy in the treatment of lower limb muscle injuries.

ELIGIBILITY:
Inclusion Criteria:

* presence of a grade III A muscle lesion of the lower limbs, according to the Mueller-Wohlfart classification, confirmed by ultrasound examination and occurred during sporting activity at least 5 days before inclusion in the study;
* no previous muscle injury in the last 6 months;
* signing of the written informed consent for participation in the study.

Exclusion Criteria:

* previous muscle injuries or bone fractures of the lower limbs in the last 6 months;
* knee instability due to previous rupture of the knee ligaments;

  • instability or previous sprain of the ankle;
* active neoplastic or infectious diseases;
* contraindications to biostimulation;
* congenital anomalies of the lower limbs.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
recovery of pain | From enrollment to 3 weeks and 3 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
Size of the lesion | From enrollment to 3 weeks and 3 months
  ultrasound evaluation of the size of the muscle lesion
Frequency of relapses | From enrollment to 3 weeks and 3 months
  Onset of new muscle injury
Return to sport activity | From enrollment to 3 months
  Number of days to return to play

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico di Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scaturro D, de Sire A, Vitagliani F, Lo Nardo D, Tomasello S, Ammendolia A, Letizia Mauro G. Effectiveness of cryo plus ultrasound therapy versus diathermy in combination with high-intensity laser therapy for pain relief in footballers with muscle injuries: A prospective study. J Back Musculoskelet Rehabil. 2024;37(3):771-780. doi: 10.3233/BMR-230265. PMID 38160343
- [Background] Medeiros DM, Aimi M, Vaz MA, Baroni BM. Effects of low-level laser therapy on hamstring strain injury rehabilitation: A randomized controlled trial. Phys Ther Sport. 2020 Mar;42:124-130. doi: 10.1016/j.ptsp.2020.01.006. Epub 2020 Jan 10. PMID 31991284
- [Background] Askling CM, Tengvar M, Tarassova O, Thorstensson A. Acute hamstring injuries in Swedish elite sprinters and jumpers: a prospective randomised controlled clinical trial comparing two rehabilitation protocols. Br J Sports Med. 2014 Apr;48(7):532-9. doi: 10.1136/bjsports-2013-093214. PMID 24620041